CLINICAL TRIAL: NCT00228215
Title: Tips for Infant and Parent Sleep (TIPS) Pilot Study
Brief Title: Tips for Infant and Parent Sleep (TIPS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Robyn Stremler, Nursing Research Associate, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1000007776
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Sleep Deprivation
Keywords: sleep; neonates; mothers; behavioural intervention
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (No Intervention)
- TIPS Intervention (Experimental)
  Interventions: Behavioral: TIPS Intervention

INTERVENTIONS:
Behavioral: TIPS Intervention — A behavioral-educational sleep intervention and support from a nurse in the immediate postpartum
  Arms: TIPS Intervention

SUMMARY:
A randomized controlled trial design will be used to answer whether a behavioral-educational sleep intervention and support from a nurse in the immediate postpartum improves maternal and infant sleep 6 weeks later.

DETAILED DESCRIPTION:
Infant and maternal sleep in the postpartum are related, and influenced by the mother's understanding of infant sleep behavior, the environmental and social cues for sleep presented to the infant, development of the infant's sleep physiology, maternal sleep habits and behaviors, and maternal feelings related to her sleep and her baby's sleep. These factors may be modifiable through the use of behavioral-educational interventions. A randomized controlled trial design will be used to answer whether a behavioral-educational sleep intervention and support from a nurse in the immediate postpartum improves maternal and infant sleep 6 weeks later. Sleep-wake patterns will be analyzed through the use of actigraphy, a wristwatch-like device that measures sleep-wake activity. This is a pilot study which will test the usefulness and practicality of this type of program, so that a larger scale study can be developed.

ELIGIBILITY:
Inclusion Criteria:

* Singleton baby born at GA >37 weeks
* baby 8 hours to 7 days old
* Mother age 16-50 years
* Normal, healthy infant as described in newborn examination
* First time parents living in the Greater Toronto Area
* Mother planning to provide fulltime care to her infant for at least the first six weeks after discharge home

Exclusion Criteria:

* Maternal or infant complications requiring prolonged hospital stay
* Previous stillbirth or neonatal death
* Maternal chronic illness
* Maternal use of medications that affect sleep (e.g. benzodiazepines, any sleep aid)
* Known drug or alcohol use beyond occasional social use
* Smoking two packs a day or more
* Either parent has a diagnosed sleep disorder (e.g. obstructive sleep apnea, narcolepsy)
* Mother's partner is working night shifts
* Mother unable to read or understand English
* No telephone in the home
* Involvement in another research protocol involving sleep

Ages: 8 Hours to 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2005-09; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Sleep outcomes (nocturnal sleep duration, total daily sleep time, time awake after sleep onset, number of night wakings, length of longest sleep periods) for women and their infants will be measured using actigraphy at 6 weeks. | 6 weeks postpartum

SECONDARY OUTCOMES:
Participant recording of sleep times, wake times, and events that occurred that might have affected sleep for the night | 6 weeks postpartum
Morning and evening fatigue measured by the Fatigue Visual Analogue Scale (Fatigue-VAS) at 6 weeks (Lee et al., 1991) | 6 weeks postpartum
Sleep disturbance measured using the General Sleep Disturbance Scale (GSDS) at both baseline and 6 weeks | 6 weeks postpartum
depressive symptomatology measured with the Edinburgh Postnatal Depression Scale (EPDS) (Cox et al., 1987)at baseline and 6 weeks | 6 weeks postpartum
levels of relatively transient, situation-related (state) anxiety as measured by the State-Trait Anxiety Inventory, state-anxiety subscale (Spielberger, 1970)at baseline and 6 weeks | 6 weeks postpartum
intervention use, perceived helpfulness of interventions, satisfaction with TIPS Pilot study involvement, and preferences for interventions and data collection methods will be assessed using a questionnaire at 6 weeks | 6 weeks postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Robyn Stremler, RN, PhD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (2):
- Canada (2):
  - The Hospital for Sick Children, Toronto, Ontario
  - Sunnybrook & Women's Health Sciences Centre - Women's College Campus, Toronto, Ontario

REFERENCES:
- [Result] Stremler R, Hodnett E, Lee K, MacMillan S, Mill C, Ongcangco L, Willan A. A behavioral-educational intervention to promote maternal and infant sleep: a pilot randomized, controlled trial. Sleep. 2006 Dec;29(12):1609-15. doi: 10.1093/sleep/29.12.1609. PMID 17252892